# Nerve block with liposomal bupivacaine yields fewer complications and similar pain relief when compared to an interscalene catheter for arthroscopic shoulder surgery: a randomized controlled trial

Principal Investigator: Amit Momaya

National Clinical Trial (NCT) Identified Number: NCT03738696

Version Number: v1.0

**06 December 2023** 

# **Table of Contents**

| S | TATI | EMEN | T OF COMPLIANCE | .1 |
|---|---|---|---|---|
| 1 | | PRO | TOCOL SUMMARY | .1 |
| | 1.1 | | Synopsis | |
| | 1.2 | | Schedule of Activities (SoA) | .2 |
| 2 | | INTR | ODUCTION | .3 |
| | 2.1 | | Study Rationale | .3 |
| | 2.2 | | Background | .3 |
| | 2.3 | | Risk/Benefit Assessment | .3 |
| | 2. | .3.1 | Known Potential Risks | .3 |
| | 2. | .3.2 | Known Potential Benefits | .3 |
| 3 | | STUE | DY DESIGN | .3 |
| | 3.1 | | Overall Design | .3 |
| | 3.2 | | End of Study Definition | .4 |
| 4 | | STUE | DY POPULATION | .4 |
| | 4.1 | | Inclusion Criteria | .4 |
| | 4.2 | | Exclusion Criteria | .4 |
| | 4.3 | | Screen Failures | .4 |
| | 4.4 | | Strategies for Recruitment and Retention | .4 |
| 5 | | STUE | DY INTERVENTION | .4 |
| | 5.1 | | Study Intervention(s) Administration Error! Bookmark not define | |
| | 5. | .1.1 | Study Intervention Description Error! Bookmark not define | d. |
| | 5. | .1.2 | Dosing and Administration Error! Bookmark not define | d. |
| 6 | | STUE | DY INTERVENTION DISCONTINUATION AND SUBJECT | |
| D | ISCO | NITNC | UATION/WITHDRAWAL | .5 |
| | 6.1 | | Discontinuation of Study Intervention | |
| | 6.2 | | Subject Discontinuation/Withdrawal from the Study | |
| | 6.3 | | Lost to Follow-Up | .5 |
| 7 | | STUE | DY ASSESSMENTS AND PROCEDURES | |
| | 7.1 | | STUDY Assessments | |
| | 7.2 | | Adverse Events and Serious Adverse Events | .6 |
| | 7. | .2.1 | Definition of Adverse Events (AE) | .6 |
| | 7. | .2.2 | Definition of Serious Adverse Events (SAE) | .6 |
| | 7. | .2.3 | Classification of an Adverse Event | .6 |
| | 7. | .2.4 | Time Period and Frequency for Event Assessment and Follow-Up | .7 |
| | 7. | .2.5 | Adverse and serious adverse Event Reporting | .8 |
| | 7.3 | | Unanticipated Problems | .8 |
| | 7. | .3.1 | Definition of Unanticipated Problems (UP) | .8 |
| | 7. | .3.2 | Unanticipated Problem Reporting | |
| 8 | | | TISTICAL CONSIDERATIONS | |
| | 8.1 | | Statistical Hypotheses | |
| | 8.2 | | Sample Size Determination | |
| | 8.3 | | Statistical Analyses | |
| | - | | | - |
| 9 | | SUPF | PORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS | ٩ |
| _ | | | | |

| 9.1 | Regulatory, Ethical, and Study Oversight Considerations | 10 |
|--------|---------------------------------------------------------|----|
| 9.1.1 | Informed Consent Process | 10 |
| 9.1.2 | Study Discontinuation and Closure | 10 |
| 9.1.3 | Confidentiality and Privacy | 11 |
| 9.1.4 | Quality Assurance and Quality Control | 11 |
| 9.1.5 | Data Handling and Record Keeping | 11 |
| 9.1.6 | Protocol Deviations | 12 |
| 9.1.7 | Conflict of Interest Policy | 12 |
| 9.2 | Abbreviations | 13 |
| 10 REF | ERENCES | 14 |

#### STATEMENT OF COMPLIANCE

The trial will be conducted in accordance with International Conference on Harmonization Good Clinical Practice (ICH GCP) and applicable United States (US) Code of Federal Regulations (CFR). The Principal Investigator will assure that no deviation from, or changes to, the protocol will take place without prior documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial subjects. All personnel involved in the conduct of this study have completed Human Subjects Protection and ICH GCP Training.

The protocol, informed consent form(s), recruitment materials, and all subject materials will be submitted to the local Institutional Review Board (IRB) for review and approval. Approval of both the protocol and the consent form must be obtained before any subject is enrolled. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented to the study. All changes to the consent form will be IRB approved; a determination will be made regarding whether a new consent needs to be obtained from subjects who provided consent, using a previously approved consent form.

#### 1 PROTOCOL SUMMARY

#### 1.1 SYNOPSIS

| Title: | Nerve block with liposomal bupivacaine yields fewer complications and similar pain relief when compared to an interscalene catheter for |
|---|---|
| | arthroscopic shoulder surgery: a randomized controlled trial |
| Study Description: | This is a blinded, randomized controlled trial to compare the control arm (continuous ropivacaine ISC) to the experimental arm (single-injection, brachial plexus nerve block using liposomal bupivacaine) in patients |
| | undergoing outpatient arthroscopic shoulder surgery at a single, tertiary academic institution. |
| Objectives: | <ul> <li>Compare complication rates</li> <li>Compare pain level, dose frequency of prescribed opioid analgesics, consumption of prescribed nonopioid analgesics, quantity and quality of sleep, and overall satisfaction with pain control</li> <li>Compare patient-reported outcome measures</li> </ul> |
| Endpoints: | <ul> <li>Patient reported complications on post-op day 0, 1, 2, 3, and 4</li> <li>Visual Analog Scale, prescribed opioid analgesic dose frequency, consumption of prescribed nonopioid analgesics, hours of uninterrupted sleep, subjective quality of sleep (0-10 scale), and pain control overall satisfaction (five-point Likert scale) on post-op day 0, 1, 2, 3, and 4</li> <li>Visual Analog Scale, Single Assessment Numeric Evaluation, American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form, and Penn Shoulder Score at 12 weeks post-op</li> </ul> |
| Study Population: | Patients greater than 19 years of age undergoing outpatient arthroscopic shoulder |
| Dhasa | Surgery Not Applicable |
| Phase: | Not Applicable |

| Description of Study | Patients in the ISC arm will have a 19 gauge Arrow Continuous Nerve Catheter |
|---|---|
| Intervention: | (Teleflex, Wayne, PA, USA) placed with a bolus of 15-20 mL of 0.5% ropivacaine given through the needle prior to threading the catheter. An elastomeric, basalonly, On-Q infusion pump (Avanos Medical, Alpharetta, GA, USA) with 0.2% ropivacaine will be started in the post-anesthesia care unit at 8 mL/hour, and the catheter will be removed by the patient after two days. For patients in the LB arm, 10 mL (133 mg) of liposomal bupivacaine (Pacira BioSciences, Parsippany, NJ, USA) mixed with 7 mL (35 mg) bolus of 0.5% bupivacaine will be injected. |
| Study Duration: | January 1, 2020 to December 1, 2021 |
| Subject Duration: | 3 months |

## 1.2 SCHEDULE OF ACTIVITIES (SOA)

- Screening/Consent Visit
- Randomization Visit
- Day of Surgery Visit
- Call 1: Evening after surgery (Day 0)
- Call 2: Day 1 morning
- Call 3: Day 1 evening
- Call 4: Day 2 morning
- Call 5: Day 2 evening
- Call 6: Day 3 morning
- Call 7: Day 3 evening
- Call 8: Day 4 morning
- Call 9: Day 4 evening

#### 2 INTRODUCTION

#### 2.1 STUDY RATIONALE

Following orthopedic surgery, patients frequently experience pain and discomfort. Multiple methods of regional anesthesia are available; however, the optimal technique to adequately manage pain while minimizing complications remains under investigation in arthroscopic shoulder surgery.

#### 2.2 BACKGROUND

After orthopaedic surgery, patients experience exquisite levels of pain due to the large, invasive and disruptive procedures performed on the musculoskeletal system. Perioperative and post-operative pain management has traditionally involved regional anesthesia, utilizing sodium-channel blockers such as bupivacaine or ropivacaine. However, their short-acting nature requires continuous infusion via an implanted catheter that remains in place for 48-72 hours. This catheter is undesirable because it can become dislodged, requires the patient to manage it, as well as return days after surgery for removal.

A modified form of bupivacaine that is bound to lipid (liposomal bupivacaine) has been shown to have a much longer duration of action than the traditional sodium channel blockers<sup>1</sup>. It is long enough that it could cover the same duration of pain as an implanted catheter and has generated interest in its potential use to control postoperative pain. Among patients undergoing total shoulder replacement, liposomal bupivacaine has shown to be non-inferior to standard catheter treatment<sup>2-6</sup>, but there is a paucity of information on its use in rotator cuff repair<sup>7</sup>. This study is meant to investigate the use of liposomal bupivacaine after arthroscopic shoulder surgery as compared to standard, catheter-infused ropivacaine.

#### 2.3 RISK/BENEFIT ASSESSMENT

#### 2.3.1 KNOWN POTENTIAL RISKS

Risks are no different than that of routine multi-modal pain control. This includes inadequate pain control, nausea, vomiting, opioid addiction, infection, headache, respiratory depression, opioid addiction, hypotension, sedation, ileus, constipation, dry mouth, and gastric ulcers.

#### 2.3.2 KNOWN POTENTIAL BENEFITS

The benefits of liposomal bupivacaine include potentially increased pain control, decreased narcotic use, and decreased catheter-associated complications including knotting and falling out. If it shows either superiority or even non-inferiority to the routine multi-modal pain management, its addition will potentially decrease adverse outcomes of current procedures.

#### 3 STUDY DESIGN

#### 3.1 OVERALL DESIGN

Patients undergoing arthroscopic shoulder surgery were prospectively assessed after randomization into either ropivacaine ISC or single-injection liposomal bupivacaine brachial plexus nerve block (LB) arms. All patients were

discharged with 5 analgesics (acetaminophen, methocarbamol, gabapentin, acetylsalicylic acid, and oxycodone) for as-needed pain relief. Preoperatively, patient demographics and baseline Visual Analog Scale, Single Assessment Numeric Evaluation, American Shoulder and Elbow Surgeons, and Penn Shoulder Scores were obtained. For the first four days postoperatively, complication rates (nausea, dyspnea, anesthetic site discomfort and/or irritation and/or leakage, and self-reported concerns and complications), pain, medication usage, and sleep data were assessed by phone survey every 12 hours. The primary outcome was overall complication rate. At 12 weeks postoperatively, Visual Analog Scale, Single Assessment Numeric Evaluation, American Shoulder and Elbow Surgeons, and Penn scores were reassessed. Outcome scores were compared with Mann-Whitney U tests, and demographics were compared with chi-squared tests. Significance was set at P < .05

#### 3.2 END OF STUDY DEFINITION

At 12 weeks postop patients will have ASES, SANE, and Penn shoulder scores calculated. This will conclude their participation in the study.

#### **4 STUDY POPULATION**

#### 4.1 INCLUSION CRITERIA

- Between ages 18 and 100 years old
- Scheduled for shoulder surgery
- Capable of providing informed consent (cognitively intact if consenting to surgery)

#### 4.2 EXCLUSION CRITERIA

- Any surgical indication other than shoulder surgery
- Any comorbidities making surgery unsafe for the patient
- Any other condition or events considered exclusionary by the PIs and/or physician Co-Is.

#### 4.3 SCREEN FAILURES

N/A

#### 4.4 STRATEGIES FOR RECRUITMENT AND RETENTION

Participants will be recruited to this study who present to the orthopaedic clinic with conditions that require arthroscopic rotator cuff repair.

#### **5 STUDY INTERVENTION**

#### 5.1 STUDY INTERVENTION DESCRIPTION

Subjects will either receive ropivacaine interscalene catheter (control group) or single shot bupivacaine interscalene block with liposomal bupivacaine interscalene block as well (study group).

#### 5.2 DOSING AND ADMINISTRATION

# 6 STUDY INTERVENTION DISCONTINUATION AND SUBJECT DISCONTINUATION/WITHDRAWAL

#### 6.1 DISCONTINUATION OF STUDY INTERVENTION

If the subject experiences adverse effects of study intervention, the intervention will be withdrawn immediately.

#### 6.2 SUBJECT DISCONTINUATION/WITHDRAWAL FROM THE STUDY

Subjects are free to withdraw from participation in the study at any time upon request.

An investigator may discontinue or withdraw a subject from the study for the following reasons:

- Significant study intervention non-compliance
- If any clinical adverse event (AE), laboratory abnormality, or other medical condition or situation occurs such that continued participation in the study would not be in the best interest of the subject

Subjects who sign the informed consent form and are randomized but do not receive the study intervention may be replaced. Subjects who sign the informed consent form, and are randomized and receive the study intervention, and subsequently withdraw, or are withdrawn or discontinued from the study, will not be replaced.

#### 6.3 LOST TO FOLLOW-UP

A subject will be considered lost to follow-up if he or she fails to return for 2 scheduled visits and is unable to be contacted by the study site staff.

The following actions must be taken if a subject fails to be available for a required study visit:

- The site will attempt to contact the subject and reschedule the missed visit and counsel the subject on the importance of maintaining the assigned visit schedule and ascertain if the subject wishes to and/or should continue in the study.
- Before a subject is deemed lost to follow-up, the investigator or designee will make every effort to regain contact with the subject (where possible, 3 telephone calls and, if necessary, a certified letter to the subject's last known mailing address or local equivalent methods). These contact attempts should be documented in the subject's medical record or study file.
- Should the subject continue to be unreachable, he or she will be considered to have withdrawn from the study with a primary reason of lost to follow-up.

#### 7 STUDY ASSESSMENTS AND PROCEDURES

#### 7.1 STUDY ASSESSMENTS

twice-daily phone calls for the first 4 days post-surgery

At each phone call, the following surveys will be performed:

- Medication Intake Survey
  - Since the last phone call:
    - Which medications have been consumed?
    - How many pills?
- Pain Survey
  - On a scale of 1-10, with 10 being the worst, what is your pain right now?
- Sleep Quality Survey
  - On a scale of 0-5, with 5 being the best, how was your sleep last night?
  - How many hours were you able to sleep before being interrupted by pain?

#### 7.2 ADVERSE EVENTS AND SERIOUS ADVERSE EVENTS

#### 7.2.1 DEFINITION OF ADVERSE EVENTS (AE)

Adverse event means any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related (21 CFR 312.32 (a)).

#### 7.2.2 DEFINITION OF SERIOUS ADVERSE EVENTS (SAE)

An adverse event (AE) is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes:

- Death
- A life-threatening adverse event (of note, the term "life-threatening" refers to an event in which the subject was at risk of death at the time of the event, rather than to an event which hypothetically might have caused death if it were more severe)
- inpatient hospitalization or prolongation of existing hospitalization
- a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- or a congenital anomaly/birth defect.

Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

#### 7.2.3 CLASSIFICATION OF AN ADVERSE EVENT

#### 7.2.3.1 SEVERITY OF EVENT

For adverse events (AEs), the following guidelines will be used to describe severity:

- **Mild** Events require minimal or no treatment and do not interfere with the subject's daily activities.
- **Moderate** Events result in a low level of inconvenience or concern with the therapeutic measures. Moderate events may cause some interference with functioning.
- **Severe** Events interrupt a subject's usual daily activity and may require systemic drug therapy or other treatment. Severe events are usually potentially life-threatening or incapacitating. Of note, the term "severe" does not necessarily equate to "serious."

#### 7.2.3.2 RELATIONSHIP TO STUDY INTERVENTION

All adverse events (AEs) must have their relationship to study intervention assessed by the clinician who examines and evaluates the subject based on temporal relationship and his/her clinical judgment. The degree of certainty about causality will be graded using the categories below. In a clinical trial, the study product must always be suspect.

- **Related** The AE is known to occur with the study intervention, there is a reasonable possibility that the study intervention caused the AE, or there is a temporal relationship between the study intervention and event. Reasonable possibility means that there is evidence to suggest a causal relationship between the study intervention and the AE.
- **Not Related** There is not a reasonable possibility that the administration of the study intervention caused the event, there is no temporal relationship between the study intervention and event onset, or an alternate etiology has been established.

#### 7.2.3.3 EXPECTEDNESS

The Principal Investigator will be responsible for determining whether an adverse event (AE) is expected or unexpected. An AE will be considered unexpected if the nature, severity, or frequency of the event is not consistent with the risk information previously described for the study intervention.

#### 7.2.4 TIME PERIOD AND FREQUENCY FOR EVENT ASSESSMENT AND FOLLOW-UP

The occurrence of an adverse event (AE) or serious adverse event (SAE) may come to the attention of study personnel during study visits and interviews of a study subject presenting for medical care, or upon review by a study monitor.

All AEs including local and systemic reactions not meeting the criteria for SAEs will be captured on the appropriate case report form (CRF). Information to be collected includes event description, time of onset, clinician's assessment of severity, relationship to study product (assessed only by those with the training and authority to make a diagnosis), and time of resolution/stabilization of the event. All AEs occurring while on study must be documented appropriately regardless of relationship. All AEs will be followed to adequate resolution.

Any medical condition that is present at the time that the subject is screened will be considered as baseline and not reported as an AE. However, if the study subject's condition deteriorates at any time during the study, it will be recorded as an AE.

Changes in the severity of an AE will be documented to allow an assessment of the duration of the event at each level of severity to be performed. AEs characterized as intermittent require documentation of onset and duration of each episode.

The Study Coordinator will record all reportable events with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation. At each study visit, the Study Coordinator will inquire about the occurrence of AE/SAEs since the last visit. Events will be followed for outcome information until resolution or stabilization.

#### 7.2.5 ADVERSE AND SERIOUS ADVERSE EVENT REPORTING

All serious adverse events must be reported to the IRB according to regulatory requirements. The Principal Investigator will immediately report to the sponsor any serious adverse event, whether or not considered study intervention related, including those listed in the protocol or package insert and must include an assessment of whether there is a reasonable possibility that the study intervention caused the event. Study endpoints that are serious adverse events (e.g., all-cause mortality) must be reported in accordance with the protocol unless there is evidence suggesting a causal relationship between the study intervention and the event (e.g., death from anaphylaxis). In that case, the investigator must immediately report the event to the sponsor.

All serious adverse events (SAEs) will be followed until satisfactory resolution or until the Principal Investigator deems the event to be chronic or the subject is stable. Other supporting documentation of the event may be requested and should be provided as soon as possible.

#### 7.3 UNANTICIPATED PROBLEMS

#### 7.3.1 DEFINITION OF UNANTICIPATED PROBLEMS (UP)

The Office for Human Research Protections (OHRP) considers unanticipated problems involving risks to subjects or others to include, in general, any incident, experience, or outcome that meets <u>all</u> of the following criteria:

- Unexpected in terms of nature, severity, or frequency given (a) the research procedures that are
  described in the protocol-related documents, such as the Institutional Review Board (IRB)approved research protocol and informed consent document; and (b) the characteristics of the
  subject population being studied;
- Related or possibly related to participation in the research ("possibly related" means there is a reasonable possibility that the incident, experience, or outcome may have been caused by the procedures involved in the research); and
- Suggests that the research places subjects or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

### 7.3.2 UNANTICIPATED PROBLEM REPORTING

The investigator will report unanticipated problems (UPs) to the reviewing Institutional Review Board (IRB). The UP report will include the following information:

- Protocol identifying information: protocol title and number, PI's name, and the IRB project number;
- A detailed description of the event, incident, experience, or outcome;
- An explanation of the basis for determining that the event, incident, experience, or outcome represents an UP;

• A description of any changes to the protocol or other corrective actions that have been taken or are proposed in response to the UP.

To satisfy the requirement for prompt reporting, UPs will be reported using the following timeline:

- UPs that are serious adverse events (SAEs) will be reported to the IRB within 10 working days of the investigator becoming aware of the event.
- Any other UP will be reported to the IRB within 10 working days of the investigator becoming aware of the problem.

#### 8 STATISTICAL CONSIDERATIONS

#### 8.1 STATISTICAL HYPOTHESES

- Primary Efficacy Endpoint(s): Postoperative Pain Scores
- Secondary Efficacy Endpoint(s): Postoperative Oral Morphine Equivalents, Analgesia Satisfaction, Analgesia Complications, Sleep Quality, and Hours of Painless Sleep

#### 8.2 SAMPLE SIZE DETERMINATION

A power analysis was conducted at 0.8 with an alpha of 0.05, using liposomal bupivacaine and ISC complication rates calculated from prior literature.

#### 8.3 STATISTICAL ANALYSES

Data analysis was performed using IBM SPSS Statistics for Macintosh, version 27 (IBM Corp., Armonk, NY, USA). Prior to study arm comparison, a Shapiro-Wilk test was performed, which indicated non-normally distributed data.

Patient age, BMI, operative time, perioperative pain scores, medication consumption, duration and quality of sleep, satisfaction, and preoperative and postoperative PROMs (VAS, SANE, ASES, and PSS) were compared using Mann-Whitney U tests.

Additional patient demographics, including gender, smokable tobacco consumption, intraoperative complications, ASA classification, CCI scores, surgical procedures, and 6 perioperative complications (nausea, dyspnea, anesthetic site discomfort and/or irritation and/or leakage, and self-reported complications), were compared with chi-squared tests. Graded measures, such as anesthetic site discomfort and irritation, were dichotomized based on severity, into "none-to-mild" and "moderate-to-severe" categories for analysis. Statistical significance was set to P < .05.

#### 9 SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

#### 9.1 REGULATORY, ETHICAL, AND STUDY OVERSIGHT CONSIDERATIONS

#### 9.1.1 INFORMED CONSENT PROCESS

#### 9.1.1.1 CONSENT/ASSENT AND OTHER INFORMATIONAL DOCUMENTS PROVIDED TO SUBJECTS

Consent forms describing in detail the study intervention, study procedures, and risks are given to the subject and written documentation of informed consent is required prior to conducting study screening procedures. A separate screening consent form will not be used.

#### 9.1.1.2 CONSENT PROCEDURES AND DOCUMENTATION

Informed consent is a process that is initiated prior to the individual's agreeing to participate in the study and continues throughout the individual's study participation. Consent forms will be Institutional Review Board (IRB)-approved and the subject will be asked to read and review the document. The investigator will explain the research study to the subject and answer any questions that may arise. A verbal explanation will be provided in terms suited to the subject's comprehension of the purposes, procedures, and potential risks of the study and of their rights as research subjects. Subjects will have the opportunity to carefully review the written consent form and ask questions prior to signing. The subjects should have the opportunity to discuss the study with their family or surrogates or think about it prior to agreeing to participate. The subject will sign the informed consent document prior to any procedures being done specifically for the study. Subjects must be informed that participation is voluntary and that they may withdraw from the study at any time, without prejudice. A copy of the informed consent document will be given to the subjects for their records. The informed consent process will be conducted and documented in the source document (including the date), and the form signed, before the subject undergoes any study-specific procedures. The rights and welfare of the subjects will be protected by emphasizing to them that the quality of their medical care will not be adversely affected if they decline to participate in this study.

#### 9.1.2 STUDY DISCONTINUATION AND CLOSURE

This study may be temporarily suspended or prematurely terminated if there is sufficient reasonable cause. Written notification, documenting the reason for study suspension or termination, will be provided by the suspending or terminating party to regulatory authorities. If the study is prematurely terminated or suspended, the Principal Investigator (PI) will promptly inform study subjects and the Institutional Review Board (IRB), will provide the reason(s) for the termination or suspension. Study subjects will be contacted, as applicable, and be informed of changes to study visit schedule.

Circumstances that may warrant termination or suspension include, but are not limited to:

- Determination of unexpected, significant, or unacceptable risk to subjects
- Demonstration of efficacy that would warrant stopping
- Insufficient compliance to protocol requirements
- Data that are not sufficiently complete and/or evaluable
- Determination that the primary endpoint has been met
- Determination of futility

Study may resume once concerns about safety, protocol compliance, and data quality are addressed, and satisfy the IRB.

#### 9.1.3 CONFIDENTIALITY AND PRIVACY

Subject confidentiality and privacy is strictly held in trust by the participating investigators and their staff. Therefore, the study protocol, documentation, data, and all other information generated will be held in strict confidence. No information concerning the study or the data will be released to any unauthorized third party without prior written approval of the Principal Investigator.

All research activities will be conducted in as private a setting as possible.

Representatives of the Institutional Review Board (IRB) may inspect all documents and records required to be maintained by the investigator, including but not limited to, medical records (office, clinic, or hospital) and pharmacy records for the subjects in this study. The clinical study site will permit access to such records.

The study subject's contact information will be securely stored at each clinical site for internal use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictated by the reviewing IRB and/or Institutional policies.

Study subject research data, which is for purposes of statistical analysis and scientific reporting, will be stored at the UAB Department of Otolaryngology research office. This will not include the subject's contact or identifying information. Rather, individual subjects and their research data will be identified by a unique study identification number. The study data entry and study management systems used by research staff will be secured and password protected.

#### 9.1.4 QUALITY ASSURANCE AND QUALITY CONTROL

The site will perform internal quality management of study conduct, data collection, documentation and completion. Quality control (QC) procedures will be completed by the Data Manager during data entry into the appropriate CRF. Any missing data or data anomalies will be communicated to the Study Coordinator for clarification/resolution.

Following written Standard Operating Procedures (SOPs), the monitors will verify that the clinical trial is conducted and data are generated are collected, documented (recorded), and reported in compliance with the protocol, International Conference on Harmonisation Good Clinical Practice (ICH GCP), and applicable regulatory requirements.

The site will provide direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and inspection by local and regulatory authorities.

#### 9.1.5 DATA HANDLING AND RECORD KEEPING

#### 9.1.5.1 DATA COLLECTION AND MANAGEMENT RESPONSIBILITIES

Data collection is the responsibility of the clinical trial staff at the site under the supervision of the Principal Investigator. The Principal Investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported.

All source documents should be completed in a neat, legible manner to ensure accurate interpretation of data.

Hard copies of source document worksheets will be used for recording data for each subject enrolled in the study. Data recorded in the case report form (CRF) derived from source documents should be consistent with the data recorded on the source documents.

#### 9.1.5.2 STUDY RECORDS RETENTION

Study documents should be retained for a minimum of 3 years after the completion of the study. These documents should be retained for a longer period, however, if required by local regulations.

#### 9.1.6 PROTOCOL DEVIATIONS

A protocol deviation is any noncompliance with the clinical trial protocol requirements. The noncompliance may be either on the part of the subject, the investigator, or the study site staff. As a result of deviations, corrective actions are to be developed by the site and implemented promptly.

These practices are consistent with ICH GCP:

- 4.5 Compliance with Protocol, sections 4.5.1, 4.5.2, and 4.5.3
- 5.1 Quality Assurance and Quality Control, section 5.1.1
- 5.20 Noncompliance, sections 5.20.1, and 5.20.2.

It is the responsibility of the Principal Investigator to use continuous vigilance to identify and report deviations within 10 working days of identification of the protocol deviation. Protocol deviations must be sent to the reviewing Institutional Review Board (IRB) per their policies. The Principal Investigator is responsible for knowing and adhering to the reviewing IRB requirements.

#### 9.1.7 CONFLICT OF INTEREST POLICY

The independence of this study from any actual or perceived influence, such as by the pharmaceutical industry, is critical. Therefore, any actual conflict of interest of persons who have a role in the design, conduct, analysis, publication, or any aspect of this trial will be disclosed and managed. Furthermore, persons who have a perceived conflict of interest will be required to have such conflicts managed in a way that is appropriate to their participation in the design and conduct of this trial.

# 9.2 ABBREVIATIONS

| AE | Adverse Event |
|---------|-----------------------------------------------------|
| ANCOVA | Analysis of Covariance |
| CFR | Code of Federal Regulations |
| CONSORT | Consolidated Standards of Reporting Trials |
| CRF | Case Report Form |
| DHHS | Department of Health and Human Services |
| GCP | Good Clinical Practice |
| HIPAA | Health Insurance Portability and Accountability Act |
| ICH | International Conference on Harmonisation |
| ICMJE | International Committee of Medical Journal Editors |
| IRB | Institutional Review Board |
| LSMEANS | Least-squares Means |
| NCT | National Clinical Trial |
| NIH | National Institutes of Health |
| OHRP | Office for Human Research Protections |
| PI | Principal Investigator |
| QA | Quality Assurance |
| QC | Quality Control |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SOA | Schedule of Activities |
| SOP | Standard Operating Procedure |
| UP | Unanticipated Problem |
| US | United States |

#### 10 REFERENCES

#### References

- 1. About Exparel: Exparel (Liposomal Bupivacaine): Pacira Bio- Sciences, Inc. 2022. Available at: https://www.exparel.com/hcp/about- exparel/exparel-liposomal-bupivacaine
- 2. Abildgaard JT, Lonergan KT, Tolan SJ, Kissenberth MJ, Hawkins RJ, Washburn R 3rd, et al. Liposomal bupivacaine versus indwelling interscalene nerve block for postoperative pain control in shoulder arthroplasty: a prospective randomized controlled trial. J Shoulder Elbow Surg 2017;26:1175-81. https://doi.org/10.1016/j.jse.2017.03.012
- 3. Administration U.S. Food & Drug. EXPAREL (Bupivacaine Liposome Injectable Suspension) Initial U.S. Approval: 1972. ORIG-1 ed2011. Accessed March 04, 2022.
- 4. Administration U.S. Food & Drug. EXPAREL (Bupivacaine Liposome Injectable Suspension) Initial U.S. Approval: 1972. SUPPL-9 ed2018. Accessed March 04, 2022.
- 5. Ali I, Gupta HO, Khazzam M, Thomas GL, Vattigunta S, Shi BY, et al. Do local liposomal bupivacaine and interscalene nerve block provide similar pain control after shoulder arthroplasty? A dual-center ran-domized controlled trial. J Shoulder Elbow Surg 2021;30(7S):S145-52. https://doi.org/10.1016/j.jse.2021.04.010
- 6. Angerame MR, Ruder JA, Odum SM, Hamid N. Pain and opioid use after total shoulder arthroplasty with injectable liposomal bupivacaine versus interscalene block. Orthopedics 2017;40:e806-11. https://doi.org/10.3928/01477447-20170608-01
- 7. Baessler AM, Moor M, Conrad DJ, Creighton J, Badman BL. Single- Shot liposomal bupivacaine reduces postoperative narcotic use following outpatient rotator cuff repair: a prospective, double-blinded, randomized controlled trial. J Bone Joint Surg Am 2020;102:1985-92. https://doi.org/10.2106/JBJS.20.00225
- 8. Ford E, Saini S, Szukics P, Assiamah AA, McMillan S. Patient-re- ported outcomes after arthroscopic shoulder surgery with interscalene brachial plexus nerve block using liposomal bupivacaine: a prospec- tive observational study. Surg Technol Int 2019;35:319-22.
- 9. Fredrickson MJ, Leightley P, Wong A, Chaddock M, Abeysekera A, Frampton C. An analysis of 1505 consecutive patients receiving contin- uous interscalene analgesia at home: a multicentre prospective safety study. Anaesthesia 2016;71:373-9. https://doi.org/10.1111/anae.13385
- 10. Hannan CV, Albrecht MJ, Petersen SA, Srikumaran U. Liposomal bupivacaine vs interscalene nerve block for pain control after shoulder arthroplasty: a retrospective cohort analysis. Am J Orthop (Belle Mead NJ) 2016;45:424-30.
- 11. Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, et al. The REDCap consortium: building an international community of software platform partners. J Biomed Inform 2019;95:103208. https://doi.org/10.1016/j.jbi.2019.103208
- 12. Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)—a metadata-driven meth- odology and workflow process for providing translational research informatics support. J Biomed Inform 2009;42:377-81. https://doi.org/
- 10.1016/j.jbi.2008.08.010